CLINICAL TRIAL: NCT00380965
Title: A Multicenter Trial Evaluating the Safety and Efficacy of Cesamet™ for the Symptomatic Treatment of Chemotherapy-Induced Neuropathic Pain in Patients With Cancer
Brief Title: Evaluation of the Efficacy of Cesamet™ for the Treatment of Pain in Patients With Chemotherapy-Induced Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NEMA Research, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB1 Study 003
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Peripheral Neuropathy; Antineoplastic Combined Chemotherapy Protocols
Keywords: Chemotherapy-induced; neuropathy; cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neoplasms | interventions — nabilone

INTERVENTIONS:
Drug: Cesamet™ (nabilone)

SUMMARY:
This study was designed to evaluate the safety and efficacy of Cesamet™ in controlling pain in subjects experiencing pain due to chemotherapy-induced neuropathic pain in patients with cancer.

DETAILED DESCRIPTION:
To determine the safety and efficacy of Cesamet™ in the symptomatic treatment of chemotherapy-induced neuropathic pain.

This is a phase IV, multicenter, open label of Cesamet™ at 1 mg daily progressing to 2mg BID in subjects with chemotherapy-induced neuropathic pain. This study has two phases: A pretreatment phase and a treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chemotherapy-induced neuropathic pain.
* Chronic daily pain present for at least 2 months.
* On stable analgesic regimen for one month.
* Baseline pain score greater than 40mm on a VAS.

Exclusion Criteria:

* Hypersensitivity to compounds in study drug or similar drugs
* Pregnant or lactating females
* Drug or alcohol abuse
* Unstable medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The Average Pain Score at target site.

SECONDARY OUTCOMES:
The Worst Pain Score at target site.
The Pain at Night Score at target site.
Quality of Life measures.
Patient satisfaction with treatment.
Safety will be assessed through the collection of AEs and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Pergolizzi, MD, Principal Investigator — NEMA Research, Inc.; Charlotte A Richmond, PhD, Study Director — NEMA Research, Inc.
Locations (2):
- United States (2):
  - South Florida Medical Research, Aventura, Florida
  - Naples Anesthesia and Pain Associates, Naples, Florida

REFERENCES:
- See also: Nema Research website — http://www.nema.net